CLINICAL TRIAL: NCT00280449
Title: Two Approaches to Providing HIV/AIDS Services in the Community to People Living With HIV/AIDS (PHAs): The Comparative Impact on Quality of Life, Access to and Expenditures for All Health and Social Services
Brief Title: Two Approaches to Providing HIV/AIDS Services in the Community to People Living With HIV/AIDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-357
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2006-01-23 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infection
Keywords: people living with HIV; quality of life
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: strengths-based case managed proactive service model

SUMMARY:
This study will examine the effects of having a case manager help PHAs access and use health, social services and practical resources that are helpful to their needs as compared to the usual more PHA self-managed approach of deciding and using services as they see necessary. New and existing users of HIV/AIDS services in Wellington-Dufferin, Waterloo and Grey-Bruce Regions who consent to this study will be randomized to receive their usual self-directed supportive, educational, medical and medical care services when they seek assistance according to their needs or these usual services augmented by case management services. They will be measured before randomization and at 3, 6 and 12 months following service use for their satisfaction with HIV/AIDS services, compliance with HIV/AIDS medication, improvement in quality of life, psychological distress, risk behaviours and expenditures for the use of a range of publicly funded services.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive individuals
* living in the community setting

Exclusion Criteria:

* cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-03; Study Completion 2007-02

PRIMARY OUTCOMES:
risk behavior, quality of life, health and social service utilization

SECONDARY OUTCOMES:
depression, satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Carvalhal, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada